CLINICAL TRIAL: NCT01617083
Title: Antibiotic Treatment Trial for the PANDAS/PANS Phenotype
Acronym: AZT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6119-128500; 270332 (Other Grant/Funding Number: Massachusetts General Hospital (MGH))
Record Dates: First submitted 2012-05-23; First posted 2012-06-12 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-03

CONDITIONS: PANS; PANDAS; Obsessive Compulsive Disorder (OCD)
Keywords: PANS; PANDAS; OCD; Tics; Azithromycin; Antibiotic Treatment
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Obsessive-Compulsive Disorder; Tics | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Active Comparator): Antibiotic used to treat infections.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Compound thickening agent with sugar and flavor additives.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Antibiotic used to treat infections
  Other Names: Zithromax; Zmax
  Arms: Azithromycin
Drug: Placebo — Thickening compound with sugar and flavoring
  Arms: Placebo

SUMMARY:
The purpose of this research study is to know if the antibiotic azithromycin, an antibiotic approved by the U.S. Food and Drug Administration (FDA) for treating infections, improves symptom severity in children with sudden and severe onset obsessive compulsive symptoms known as PANS, Pediatric Acute Onset Neuropsychiatric Syndrome, and PANDAS, Pediatric Autoimmune Neuropsychiatric Disorder Associated with Streptococcus. This study seeks to compare the effects of placebo vs. azithromycin on Obsessive Compulsive Disorder (OCD) symptom severity as well as to assess immune risk factors in children with PANDAS/PANS. Obsessions are repetitive, unwanted thoughts or worries that may be unpleasant, silly, or embarrassing. Compulsions are repetitive or ritualistic actions that are performed to ease anxiety or worries. Doctors think these symptoms may be caused or exacerbated by certain infections such as Streptococcus pyogenes, Mycoplasma pneumonia, Borrelia burgordfi, etc. These infections commonly cause strep throat, walking pneumonia, and Lyme Disease, among others.

This study will involve a 4 week double-blind, placebo-controlled randomized trial of azithromycin (Double Blind Phase). At the end of this 4 week trial, the child will be assigned to azithromycin for 8 weeks (Open Label Phase). At the end of these 12 weeks, a Naturalistic Observation phase will assess the child's symptom characteristics for up to 40 weeks.

The study hypothesizes that children receiving antibiotic will show significantly greater overall improvement in severity compared with placebo, and that children with sudden onset of OCD and whose subsequent course shows dramatic fluctuations will have evidence of immune risk factors that predisposes to this presentation.

DETAILED DESCRIPTION:
Accumulating evidence suggests that a subset of children with obsessive compulsive disorder (OCD) have a symptom course that is temporally associated with infections (group A Streptococcus, Mycoplasma, Borrelia burgordfi, etc.). The intent of this proposal is to test the hypotheses that: 1) this subset of children with OCD known as Pediatric Acute Onset Neuropsychiatric Syndrome (PANS) and the specific subset associated with Streptococcus, PANDAS (Pediatric Autoimmune Neuropsychiatric Disorder Associated with Streptococcus), experience symptom onset and exacerbations due to autoimmune/inflammatory responses to infectious triggers and, 2) antibiotic treatment will reduce symptom severity. Investigators have reported improvement in neuropsychiatric symptoms of patients presenting with PANDAS following antibiotic treatment (Murphy & Pichichero, 2002; Snider, Lougee, Slattery et al., 2005). Difficulties with study design and small sample size of early antibiotic trials limit the influence of their findings (Kurlan & Kaplan, 2004) although anecdotally, many families report often dramatic improvements in OCD symptoms after antibiotic therapy.

The proposed study is a 4 week double-blind placebo-controlled study of the efficacy of azithromycin once daily on OCD symptom severity in children ages 4-14 years presenting with the PANS phenotype. An 8 week open label phase will be offered to all subjects completing the 1-month trial to assess longer term efficacy and tolerability (12 weeks total antibiotics for those on active, 8 weeks for those on placebo). At the end of week 8, the child can transition to best clinical care practice (cognitive behavioral therapy, additional medication trials, etc) if not fully remitted. The rate and timing of any relapse will be assessed but are not the primary outcome variables. Evaluations will consist of: 1) semi-structured psychiatric diagnostic interviews and rating scales to establish psychiatric diagnoses and monitor severity of psychiatric symptoms, particularly obsessive compulsive behavior and tics; 2) parent and child-report questionnaires to elicit information regarding infections and clinical correlates of PANS attributes; 3) physical and neurological examinations; and 4) laboratory studies.

Aim 1: To compare, in randomized controlled fashion, placebo vs. antibiotic on changes in overall symptom severity for obsessive-compulsive symptoms among children with PANS phenotype. Changes from baseline and clinical status at end of study will be compared for the study arms. Primary endpoint will be change on the Children's Yale Brown Obsessive Compulsive scale (CY-BOCS). Secondary measures of interest include severity and improvement measures on the Clinical Global Impression Severity/Improvement scale, quality of life measures, and weekly ratings of mood, anxiety, attention deficit hyperactivity and tic symptoms. Hypothesis: Children receiving antibiotic will show significantly greater overall improvement in severity compared with placebo. Children that meet PANDAS/PANS criteria and have current OCD symptoms of less than 6 months duration will be enrolled in a double-blind placebo-controlled randomized trial of azithromycin for 4 weeks. Subjects will be followed weekly during the 3 months (4-week antibiotic treatment trial, 8 weeks open label treatment). Although earlier trials have had mixed results, these studies have primarily enrolled subjects with longer illness durations and used traditional prophylactic doses in contrast to the standard treatment dose of this study. Since treatment doses of antibiotic decrease antigenic load, one can speculate that treatment level doses, rather than prophylactic doses, may best attenuate neuropsychiatric sequelae. Secondary neuromodulating or immune modulating properties at higher dose of antibiotics may also be a possible mode of therapeutic action. The timing of treatment response and moderators and predictors of response will also be assessed.

Aim 2: To assess immune risk factors in children with PANDAS/PANS. The data and biological specimens (blood, cultures, etc) for all subjects consented for Aim 1 will, be entered into a database and repository to assess further these clinical phenotypes. Subjects that do not qualify for randomization (medication allergy or current long term antibiotic therapy) or decline randomization (e.g. travel required for future visits) will be permitted to contribute to Aim 2, i.e. collection of baseline symptom severity and immune marker assessment. Hypothesis: It is hypothesized that children with sudden onset of OCD and whose subsequent course shows dramatic fluctuations will have evidence of immune risk factors that predisposes to this presentation. Certain subject characteristics such as age, duration of illness, characteristics of exacerbation episodes, type and number of prior infections, and co-occurring disorders may influence treatment response. Immunologic markers that may help with determining pathobiology and treatment response will be explored including pathogen detection array to identify potential infectious triggers, cytokine array to explore inflammatory processes and specific antibody assay to assess potential mediators. In order to differentiate those children that may most benefit from antibiotic prophylaxis from those that do not benefit, analytic strategies to refine an antibiotic-responsive phenotype will be explored.

Rationale: Based on the PI's observations from research and clinical patients being referred for PANDAS (60 patients per year), patients have had most improvement when higher doses of antibiotics are used, often relapsing on prophylactic doses. The best response rates have been antibiotics designed to treat beta lactamase co-pathogens such as azithromycin, cephalosporins or amoxicillin/clavulanic acid. Observed response rates are typically within 3 weeks although some subjects appear to take longer to gain response. These observations deserve further study. Azithromycin was chosen due to improved tolerance, once daily dosing regimen, coverage against other microbes implicated in PANS and low risk for allergic reaction or exclusion.

Randomization: Study medication and matching placebo will be provided by the research pharmacy. Some of the services provided will include blinding of study drug, packaging and labeling, and randomization. Subjects who are randomized will receive either antibiotic or placebo in a 1:1 ratio. Both investigator and study participant will be blinded to the treatment assignment. Randomization will not be revealed to the investigator or the study participants until all participants have completed the study or in the event of serious adverse event (SAE).

Dosing: Azithromycin or placebo every 24 hours will be dispensed. Antibiotic will be transferred to identical bottles as placebo and dispensed without the manufacturer label. Labels will be identical with matching dose volumes for each. Flavor, color and texture will be matched to best of ability. Participants and parents will be instructed to not discuss the actual medication with anyone in the study team except the designated person dispensing the medication.

Study participation is entirely voluntary. If at any time a participant wishes to discontinue the use of study medication, they can notify the study coordinator and if the family is willing, they can choose to enter the naturalistic phase or discontinue the study.

Naturalistic Observation Phase: After the subject's completion of the active phase of the study (baseline to end of week 12 as determined by subject eligibility, medication tolerance, etc), the family will be given the choice to opt in or opt out of a naturalistic follow up on a monthly basis until end of week 52. The family will be provided a monthly PANS scale and questionnaire regarding the child's current treatment. Depending on which option works best for them, they can return by the forms by mail or complete online.

Compliance Monitoring: Azithromycin, with daily dosing, has higher rates of adherence than other antibiotics with more frequent dosing. The parent of the child will be educated about optimal dosing and compliance. Each unit dose will be labeled specifically with the participants identification number. The clinical coordinator will document each batch of medication on the dispensing log. Each batch of study medication will include supply until next scheduled visit plus one week to cover any difficulty returning to study in the scheduled interval. All study medication will be accounted for throughout the study by the investigator or the designee.

End of Treatment Alternatives: Standard of care treatment options are unavailable for the initial 8 weeks, after which point families will have multiple options for post-study care if needed. Until better guidelines are developed, children in the PANDAS/PANS subgroup should also be given the chance to benefit from evidence based treatments that may lessen the severity of a future flare up. From our previous work (Storch, Murphy, Geffken et al., 2006), we believe that remaining OCD symptoms are best treated with CBT unless the child is still too severe to engage in therapy. CBT can help children remodel automatic responses to obsessions, teach skills that should prove helpful if symptoms do recur and also help families with behavioral strategies to lessen the risk of disrupted functioning and accommodation. Children often report feeling empowered from coping, relaxation, and resiliency skills learned in cognitive behavioral therapy (CBT). Antidepressants approved for OCD are an option to consider for those that appear to have a chronic stable course but many youth with a PANS presentation are incapacitated by these sudden and severe symptoms, with many parents feeling too desperate (Murphy, observations) to wait the typical 10-12 weeks for SSRIs to achieve full efficacy. Many of these children are highly sensitive to usual starting doses (Murphy, Storch, & Strawser, 2006) but do well when started on a low dose (e.g. sertraline at 6.25mg) and gradually increased as tolerated. Patients with tics respond well to a variety of evidence based pharmacologic agents and behavioral treatments if needed due to symptom severity and impairment. Following the study all subjects with incomplete remission will be referred for CBT in the outpatient clinics or the community based on parent preference. The investigative team has considerable experience in the application of this approach for pediatric OCD (Murphy et al., 2007) and collaborates closely with outpatient providers.

Adverse effects: Every effort should be made to identify prior history of adverse effects to antibiotics prior to the randomization phase (exclusion criterion). In the event of Candidiasis, other opportunistic overgrowth or allergic reaction, the recommendations by the primary care physician (PCP) of the child will be followed. As this adverse event is unlikely except during treatment with antibiotics, blinding will be compromised and the child will be considered a drop due to adverse event. Open label probiotics will be provided to subjects in both study arms in all phases to be taken daily. In the event of an SAE, the blind should be broken only if knowing the treatment status is of significance to the course of treatment. If at any time the blinding becomes otherwise compromised, the subject will exit the randomized control trial (RCT) portion of the study. The date, time, and reason or situation surrounding unblinding must be documented as completely as possible. All SAEs should also be reported to the institutional review board (IRB) as soon as possible. Laboratory tests (CBC, metabolic panel, urine toxicology and pregnancy test [for post-pubescent females]) and an EKG will be obtained at baseline. Every 2 weeks, liver function testing will be done to monitor for hepatic toxicity risks as well as an EKG to monitor for cardiac risks (increased QTc).

ELIGIBILITY:
Inclusion Criteria:

* Ages 4 -14 years.
* Presence of OCD and at least two of the following:

  1. Anxieties e.g. new onset separation anxiety
  2. Sensory abnormalities (tactile/auditory/visual defensiveness or visual misperceptions)
  3. Behavioral Regression (e.g. new onset impulsivity, hyperactivity, meltdowns)
  4. Deterioration in school performance or in handwriting
  5. Emotional lability and/or depression
  6. Urinary symptoms (frequent urination or enuresis)
  7. Sleep disturbances Anorexia
* Current episode OCD of recent onset (less or equal to 6 months) associated with infection
* Symptom onset appears temporally related to infection or exposure
* Symptoms are of moderate severity with significant impairment (CGI of moderate or worse) and CY-BOCS of more or equal to 16.
* Parental willingness to accompany their child for multiple study visits and be responsible for medication compliance.

Exclusion Criteria:

* History of Rheumatic Fever including Sydenham's Chorea (heart murmur, frank chorea, EKG PR or QTc prolongation, abnormal reflexes (Gordon-Hey reflex)).
* Diagnosis of autism (moderate - severe), schizophrenia, mental retardation or chronic degenerative neurological disease.
* Any illness for which antibiotic treatment may be contraindicated (e.g. Liver disease).
* Personal history of adverse reaction or allergy to azithromycin.
* Recent or planned psychopharmacologic (4 weeks for most medications or 8 weeks for SSRIs) treatment changes.
* Antibiotic prophylaxis therapy or history of neuropsychiatric non-response to prior antibiotic trial.
* Currently participating in cognitive behavioral therapy or habit reversal therapy for OCD and/or tics.
* Weight less than 15 kilograms
* Concurrent therapy with medications that may increase adverse effects (eg. pimozide, citalopram, tricyclic antidepressants, etc).

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Murphy, MD, Principal Investigator — University of South Florida
Locations (1):
- Rothman Center for Neuropsychiatry, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen AJ, Leonard HL, Swedo SE. Case study: a new infection-triggered, autoimmune subtype of pediatric OCD and Tourette's syndrome. J Am Acad Child Adolesc Psychiatry. 1995 Mar;34(3):307-11. doi: 10.1097/00004583-199503000-00015. PMID 7896671
- [Background] Chia KS. Multivariate statistical analysis: a brief introduction. Ann Acad Med Singap. 1999 Nov;28(6):879-80. No abstract available. PMID 10672410
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430
- [Background] Bronze MS, Dale JB. Epitopes of streptococcal M proteins that evoke antibodies that cross-react with human brain. J Immunol. 1993 Sep 1;151(5):2820-8. PMID 7689617
- [Background] Brook I. The role of beta-lactamase-producing bacteria in the persistence of streptococcal tonsillar infection. Rev Infect Dis. 1984 Sep-Oct;6(5):601-7. doi: 10.1093/clinids/6.5.601. PMID 6390637
- [Background] Brook I. Failure of penicillin to eradicate group A beta-hemolytic streptococci tonsillitis: causes and management. J Otolaryngol. 2001 Dec;30(6):324-9. doi: 10.2310/7070.2001.19359. PMID 11771001
- [Background] Brook I. The role of beta-lactamase producing bacteria and bacterial interference in streptococcal tonsillitis. Int J Antimicrob Agents. 2001 Jun;17(6):439-42. doi: 10.1016/s0924-8579(01)00321-1. PMID 11397612
- [Background] Brook I. A pooled comparison of cefdinir and penicillin in the treatment of group a beta-hemolytic streptococcal pharyngotonsillitis. Clin Ther. 2005 Aug;27(8):1266-73. doi: 10.1016/j.clinthera.2005.08.003. PMID 16199251
- [Background] Brook I, Dohar JE. Management of group A beta-hemolytic streptococcal pharyngotonsillitis in children. J Fam Pract. 2006 Dec;55(12):S1-11; quiz S12. PMID 17137534
- [Background] Brooks-Gunn J, Warren MP, Rosso J, Gargiulo J. Validity of self-report measures of girls' pubertal status. Child Dev. 1987 Jun;58(3):829-41. PMID 3608653
- [Background] Brooks BM, Hart CA, Coleman JW. Differential effects of beta-lactams on human IFN-gamma activity. J Antimicrob Chemother. 2005 Dec;56(6):1122-5. doi: 10.1093/jac/dki373. Epub 2005 Oct 20. PMID 16239287
- [Background] Brooks BM, Thomas AL, Coleman JW. Benzylpenicillin differentially conjugates to IFN-gamma, TNF-alpha, IL-1beta, IL-4 and IL-13 but selectively reduces IFN-gamma activity. Clin Exp Immunol. 2003 Feb;131(2):268-74. doi: 10.1046/j.1365-2249.2003.02069.x. PMID 12562387
- [Background] Budman CL, Kerjakovic M, Bruun RD. Viral infection and tic exacerbation. J Am Acad Child Adolesc Psychiatry. 1997 Feb;36(2):162. doi: 10.1097/00004583-199702000-00004. No abstract available. PMID 9031566
- [Background] Carapetis JR, Currie BJ. Rheumatic chorea in northern Australia: a clinical and epidemiological study. Arch Dis Child. 1999 Apr;80(4):353-8. doi: 10.1136/adc.80.4.353. PMID 10086943
- [Background] Cardona F, Orefici G. Group A streptococcal infections and tic disorders in an Italian pediatric population. J Pediatr. 2001 Jan;138(1):71-5. doi: 10.1067/mpd.2001.110325. PMID 11148515
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Constantino, J., & CP, G. The Social Responsiveness Scale (SRS) Manual. Los Angeles: Western Psychological Services, 2005.
- [Background] Cook EH, Wagner KD, March JS, Biederman J, Landau P, Wolkow R, Messig M. Long-term sertraline treatment of children and adolescents with obsessive-compulsive disorder. J Am Acad Child Adolesc Psychiatry. 2001 Oct;40(10):1175-81. doi: 10.1097/00004583-200110000-00011. PMID 11589530
- [Background] Currie BJ. Are the currently recommended doses of benzathine penicillin G adequate for secondary prophylaxis of rheumatic fever? Pediatrics. 1996 Jun;97(6 Pt 2):989-91. PMID 8637788
- [Background] Dajani A, Taubert K, Ferrieri P, Peter G, Shulman S. Treatment of acute streptococcal pharyngitis and prevention of rheumatic fever: a statement for health professionals. Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, the American Heart Association. Pediatrics. 1995 Oct;96(4 Pt 1):758-64. PMID 7567345
- [Background] Diggle, P. Analysis of longitudinal data. Oxford University Press, 2002.
- [Background] Garvey MA, Perlmutter SJ, Allen AJ, Hamburger S, Lougee L, Leonard HL, Witowski ME, Dubbert B, Swedo SE. A pilot study of penicillin prophylaxis for neuropsychiatric exacerbations triggered by streptococcal infections. Biol Psychiatry. 1999 Jun 15;45(12):1564-71. doi: 10.1016/s0006-3223(99)00020-7. PMID 10376116
- [Background] Garvey MA, Swedo SE. Sydenham's chorea. Clinical and therapeutic update. Adv Exp Med Biol. 1997;418:115-20. doi: 10.1007/978-1-4899-1825-3_28. No abstract available. PMID 9331612
- [Background] Gerson AC, Gerring JP, Freund L, Joshi PT, Capozzoli J, Brady K, Denckla MB. The Children's Affective Lability Scale: a psychometric evaluation of reliability. Psychiatry Res. 1996 Dec 20;65(3):189-98. doi: 10.1016/s0165-1781(96)02851-x. PMID 9029668
- [Background] Gioia GA, Isquith PK, Retzlaff PD, Espy KA. Confirmatory factor analysis of the Behavior Rating Inventory of Executive Function (BRIEF) in a clinical sample. Child Neuropsychol. 2002 Dec;8(4):249-57. doi: 10.1076/chin.8.4.249.13513. PMID 12759822
- [Background] Giulino L, Gammon P, Sullivan K, Franklin M, Foa E, Maid R, March JS. Is parental report of upper respiratory infection at the onset of obsessive-compulsive disorder suggestive of pediatric autoimmune neuropsychiatric disorder associated with streptococcal infection? J Child Adolesc Psychopharmacol. 2002 Summer;12(2):157-64. doi: 10.1089/104454602760219199. PMID 12188984
- [Background] Green B, Shirk S, Hanze D, Wanstrath J. The Children's Global Assessment Scale in clinical practice: an empirical evaluation. J Am Acad Child Adolesc Psychiatry. 1994 Oct;33(8):1158-64. doi: 10.1097/00004583-199410000-00011. PMID 7982866
- [Background] Guchev IA, Klochkov OI, Ivanitsa GV, Pervov IuA, Shturmina SM, Rosman SV. [Efficacy and safety of azithromycin prophylaxis of respiratory tract infections in military community]. Antibiot Khimioter. 2004;49(8-9):34-5, 37-42. Russian. PMID 15727144
- [Background] Guilherme L, Kalil J, Cunningham M. Molecular mimicry in the autoimmune pathogenesis of rheumatic heart disease. Autoimmunity. 2006 Feb;39(1):31-9. doi: 10.1080/08916930500484674. PMID 16455580
- [Background] Guy, W. Assessment Manual for Psychopharmacology, rev. edn. Rockville, MD: National Institute of Mental Health, 1976.
- [Background] Hagelskjaer LH, Hansen NJ. [Neurological complications of Mycoplasma pneumoniae infections]. Ugeskr Laeger. 1993 Apr 26;155(17):1265-9. Danish. PMID 8506572
- [Background] Hamstra-Bletz L, Blote AW. A longitudinal study on dysgraphic handwriting in primary school. J Learn Disabil. 1993 Dec;26(10):689-99. doi: 10.1177/002221949302601007. PMID 8151209
- [Background] Husby G, van de Rijn I, Zabriskie JB, Abdin ZH, Williams RC Jr. Antibodies reacting with cytoplasm of subthalamic and caudate nuclei neurons in chorea and acute rheumatic fever. J Exp Med. 1976 Oct 1;144(4):1094-110. doi: 10.1084/jem.144.4.1094. PMID 789810
- [Background] Jacobs MR, Johnson CE. Macrolide resistance: an increasing concern for treatment failure in children. Pediatr Infect Dis J. 2003 Aug;22(8 Suppl):S131-8. doi: 10.1097/00006454-200308001-00004. PMID 14566999
- [Background] Kantor L, Hewlett GH, Gnegy ME. Enhanced amphetamine- and K+-mediated dopamine release in rat striatum after repeated amphetamine: differential requirements for Ca2+- and calmodulin-dependent phosphorylation and synaptic vesicles. J Neurosci. 1999 May 15;19(10):3801-8. doi: 10.1523/JNEUROSCI.19-10-03801.1999. PMID 10234012
- [Background] Karno M, Golding JM, Sorenson SB, Burnam MA. The epidemiology of obsessive-compulsive disorder in five US communities. Arch Gen Psychiatry. 1988 Dec;45(12):1094-9. doi: 10.1001/archpsyc.1988.01800360042006. PMID 3264144
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Kerbeshian J, Burd L, Pettit R. A possible post-streptococcal movement disorder with chorea and tics. Dev Med Child Neurol. 1990 Jul;32(7):642-4. PMID 2391015
- [Background] Khanna S, Ravi V, Shenoy PK, Chandramuki A, Channabasavanna SM. Cerebrospinal fluid viral antibodies in obsessive-compulsive disorder in an Indian population. Biol Psychiatry. 1997 Apr 15;41(8):883-90. doi: 10.1016/S0006-3223(96)00174-6. PMID 9099415
- [Background] Kiessling LS, Marcotte AC, Culpepper L. Antineuronal antibodies: tics and obsessive-compulsive symptoms. J Dev Behav Pediatr. 1994 Dec;15(6):421-5. PMID 7884013
- [Background] Kirvan CA, Swedo SE, Heuser JS, Cunningham MW. Mimicry and autoantibody-mediated neuronal cell signaling in Sydenham chorea. Nat Med. 2003 Jul;9(7):914-20. doi: 10.1038/nm892. PMID 12819778
- [Background] Kirvan CA, Swedo SE, Kurahara D, Cunningham MW. Streptococcal mimicry and antibody-mediated cell signaling in the pathogenesis of Sydenham's chorea. Autoimmunity. 2006 Feb;39(1):21-9. doi: 10.1080/08916930500484757. PMID 16455579
- [Background] Kirvan CA, Swedo SE, Snider LA, Cunningham MW. Antibody-mediated neuronal cell signaling in behavior and movement disorders. J Neuroimmunol. 2006 Oct;179(1-2):173-9. doi: 10.1016/j.jneuroim.2006.06.017. Epub 2006 Jul 27. PMID 16875742
- [Background] Kurlan R, Kaplan EL. The pediatric autoimmune neuropsychiatric disorders associated with streptococcal infection (PANDAS) etiology for tics and obsessive-compulsive symptoms: hypothesis or entity? Practical considerations for the clinician. Pediatrics. 2004 Apr;113(4):883-6. doi: 10.1542/peds.113.4.883. PMID 15060240
- [Background] Kushner HI, Kiessling LS. The controversy over the classification of Gilles de la Tourette's syndrome, 1800-1995. Perspect Biol Med. 1996 Spring;39(3):409-35. doi: 10.1353/pbm.1996.0010. No abstract available. PMID 8657554
- [Background] Landgraf, J. M., Abetz, L., & Ware, J. E. The CHQ user's manual. Boston: The Health Institute, New England Medical Center, 1996.
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Leckman JF, Sholomskas D, Thompson WD, Belanger A, Weissman MM. Best estimate of lifetime psychiatric diagnosis: a methodological study. Arch Gen Psychiatry. 1982 Aug;39(8):879-83. doi: 10.1001/archpsyc.1982.04290080001001. PMID 7103676
- [Background] Leonard HL, Swedo SE, Rapoport JL, Rickler KC, Topol D, Lee S, Rettew D. Tourette syndrome and obsessive-compulsive disorder. Adv Neurol. 1992;58:83-93. No abstract available. PMID 1414648
- [Background] Lewin AB, Storch EA, Mutch PJ, Murphy TK. Neurocognitive functioning in youth with pediatric autoimmune neuropsychiatric disorders associated with streptococcus. J Neuropsychiatry Clin Neurosci. 2011 Fall;23(4):391-8. doi: 10.1176/jnp.23.4.jnp391. PMID 22231309
- [Background] Lunsing RJ, Hadders-Algra M, Huisjes HJ, Touwen BC. Minor neurological dysfunction from birth to 12 years. I: Increase during late school-age. Dev Med Child Neurol. 1992 May;34(5):399-403. doi: 10.1111/j.1469-8749.1992.tb11451.x. PMID 1375566
- [Background] Mahone EM, Cirino PT, Cutting LE, Cerrone PM, Hagelthorn KM, Hiemenz JR, Singer HS, Denckla MB. Validity of the behavior rating inventory of executive function in children with ADHD and/or Tourette syndrome. Arch Clin Neuropsychol. 2002 Oct;17(7):643-62. PMID 14591848
- [Background] Matza LS, Rentz AM, Secnik K, Swensen AR, Revicki DA, Michelson D, Spencer T, Newcorn JH, Kratochvil CJ. The link between health-related quality of life and clinical symptoms among children with attention-deficit hyperactivity disorder. J Dev Behav Pediatr. 2004 Jun;25(3):166-74. doi: 10.1097/00004703-200406000-00005. PMID 15194901
- [Background] Mell LK, Davis RL, Owens D. Association between streptococcal infection and obsessive-compulsive disorder, Tourette's syndrome, and tic disorder. Pediatrics. 2005 Jul;116(1):56-60. doi: 10.1542/peds.2004-2058. PMID 15995031
- [Background] Meyers, J., & Meyers, K. Rey Complex Figure Test and recognition trial: Professional manual. Psychological Assessment Resources, 1995.
- [Background] Miettinen M, Matikainen S, Vuopio-Varkila J, Pirhonen J, Varkila K, Kurimoto M, Julkunen I. Lactobacilli and streptococci induce interleukin-12 (IL-12), IL-18, and gamma interferon production in human peripheral blood mononuclear cells. Infect Immun. 1998 Dec;66(12):6058-62. doi: 10.1128/IAI.66.12.6058-6062.1998. PMID 9826398
- [Background] MILLER JM, STANCER SL, MASSELL BF. A controlled study of beta hemolytic streptococcal infection in rheumatic families. II. Penicillin prophylaxis among rheumatic fever subjects, comparing different regimens. Am J Med. 1958 Dec;25(6):845-56. doi: 10.1016/0002-9343(58)90057-3. No abstract available. PMID 13606137
- [Background] Mineur YS, Picciotto MR, Sanacora G. Antidepressant-like effects of ceftriaxone in male C57BL/6J mice. Biol Psychiatry. 2007 Jan 15;61(2):250-2. doi: 10.1016/j.biopsych.2006.04.037. Epub 2006 Jul 24. PMID 16860779
- [Background] Morikawa K, Torii I, Morikawa S. Modulation of IgD and CD20 by ligation of CD5 on tonsillar B cells. Scand J Immunol. 2002 Jan;55(1):44-52. doi: 10.1046/j.1365-3083.2002.00987.x. PMID 11841691
- [Background] Muller N, Riedel M, Forderreuther S, Blendinger C, Abele-Horn M. Tourette's syndrome and mycoplasma pneumoniae infection. Am J Psychiatry. 2000 Mar;157(3):481-2. doi: 10.1176/appi.ajp.157.3.481-a. No abstract available. PMID 10698843
- [Background] Muller N, Riedel M, Blendinger C, Oberle K, Jacobs E, Abele-Horn M. Mycoplasma pneumoniae infection and Tourette's syndrome. Psychiatry Res. 2004 Dec 15;129(2):119-25. doi: 10.1016/j.psychres.2004.04.009. PMID 15590039
- [Background] Murphy BS, Sundareshan V, Cory TJ, Hayes D Jr, Anstead MI, Feola DJ. Azithromycin alters macrophage phenotype. J Antimicrob Chemother. 2008 Mar;61(3):554-60. doi: 10.1093/jac/dkn007. Epub 2008 Jan 29. PMID 18230686
- [Background] Murphy ML, Pichichero ME. Prospective identification and treatment of children with pediatric autoimmune neuropsychiatric disorder associated with group A streptococcal infection (PANDAS). Arch Pediatr Adolesc Med. 2002 Apr;156(4):356-61. doi: 10.1001/archpedi.156.4.356. PMID 11929370
- [Background] Murphy TK, Sajid M, Soto O, Shapira N, Edge P, Yang M, Lewis MH, Goodman WK. Detecting pediatric autoimmune neuropsychiatric disorders associated with streptococcus in children with obsessive-compulsive disorder and tics. Biol Psychiatry. 2004 Jan 1;55(1):61-8. doi: 10.1016/s0006-3223(03)00704-2. PMID 14706426
- [Background] Murphy TK, Snider LA, Mutch PJ, Harden E, Zaytoun A, Edge PJ, Storch EA, Yang MC, Mann G, Goodman WK, Swedo SE. Relationship of movements and behaviors to Group A Streptococcus infections in elementary school children. Biol Psychiatry. 2007 Feb 1;61(3):279-84. doi: 10.1016/j.biopsych.2006.08.031. Epub 2006 Nov 27. PMID 17126304
- [Background] Murphy TK, Storch EA, Lewin AB, Edge PJ, Goodman WK. Clinical factors associated with pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections. J Pediatr. 2012 Feb;160(2):314-9. doi: 10.1016/j.jpeds.2011.07.012. Epub 2011 Aug 25. PMID 21868033
- [Background] Murphy, T. K., Storch, E. A., & Strawser, M. S. Case Report: Selective Serotonin Reuptake Inhibitor-Induced Behavioral Activation in the PANDAS Subtype. [case report]. Primary Psychiatry, 13(8), 87-89, 2006.
- [Background] Murr C, Gerlach D, Widner B, Dierich MP, Fuchs D. Neopterin production and tryptophan degradation in humans infected by Streptococcus pyogenes. Med Microbiol Immunol. 2001 Apr;189(3):161-3. doi: 10.1007/s430-001-8023-3. PMID 11388614
- [Background] O'Connell PJ, Wang X, Leon-Ponte M, Griffiths C, Pingle SC, Ahern GP. A novel form of immune signaling revealed by transmission of the inflammatory mediator serotonin between dendritic cells and T cells. Blood. 2006 Feb 1;107(3):1010-7. doi: 10.1182/blood-2005-07-2903. Epub 2005 Oct 13. PMID 16223770
- [Background] Perlmutter SJ, Garvey MA, Castellanos X, Mittleman BB, Giedd J, Rapoport JL, Swedo SE. A case of pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections. Am J Psychiatry. 1998 Nov;155(11):1592-8. doi: 10.1176/ajp.155.11.1592. No abstract available. PMID 9812123
- [Background] Perwien AR, Faries DE, Kratochvil CJ, Sumner CR, Kelsey DK, Allen AJ. Improvement in health-related quality of life in children with ADHD: an analysis of placebo controlled studies of atomoxetine. J Dev Behav Pediatr. 2004 Aug;25(4):264-71. doi: 10.1097/00004703-200408000-00006. PMID 15308927
- [Background] Piacentini J, Bergman RL, Keller M, McCracken J. Functional impairment in children and adolescents with obsessive-compulsive disorder. J Child Adolesc Psychopharmacol. 2003;13 Suppl 1:S61-9. doi: 10.1089/104454603322126359. PMID 12880501
- [Background] Piacentini, J. C., & Jaffer, M. P., J. C., & Jaffer, M. Measuring functional impairment in youngsters with OCD: Manual for the Child OCD Impact Scale (COIS). Los Angeles, UCLA Department of Psychiatry, 1999.
- [Background] Pichichero ME, Casey JR, Mayes T, Francis AB, Marsocci SM, Murphy AM, Hoeger W. Penicillin failure in streptococcal tonsillopharyngitis: causes and remedies. Pediatr Infect Dis J. 2000 Sep;19(9):917-23. doi: 10.1097/00006454-200009000-00035. PMID 11001127
- [Background] Pichichero ME, Gooch WM 3rd. Comparison of cefdinir and penicillin V in the treatment of pediatric streptococcal tonsillopharyngitis. Pediatr Infect Dis J. 2000 Dec;19(12 Suppl):S171-3. doi: 10.1097/00006454-200012001-00007. PMID 11144400
- [Background] Pittenger C, Krystal JH, Coric V. Glutamate-modulating drugs as novel pharmacotherapeutic agents in the treatment of obsessive-compulsive disorder. NeuroRx. 2006 Jan;3(1):69-81. doi: 10.1016/j.nurx.2005.12.006. PMID 16490414
- [Background] PRECHTL HF, STEMMER J. The choreiform syndrome in children. Dev Med Child Neurol. 1962 Apr;4:119-27. doi: 10.1111/j.1469-8749.1962.tb03120.x. No abstract available. PMID 14488567
- [Background] Rentz AM, Matza LS, Secnik K, Swensen A, Revicki DA. Psychometric validation of the child health questionnaire (CHQ) in a sample of children and adolescents with attention-deficit/hyperactivity disorder. Qual Life Res. 2005 Apr;14(3):719-34. doi: 10.1007/s11136-004-0832-9. PMID 16022065
- [Background] Richter SS, Heilmann KP, Beekmann SE, Miller NJ, Miller AL, Rice CL, Doern CD, Reid SD, Doern GV. Macrolide-resistant Streptococcus pyogenes in the United States, 2002-2003. Clin Infect Dis. 2005 Sep 1;41(5):599-608. doi: 10.1086/432473. PMID 16080080
- [Background] Rothstein JD, Patel S, Regan MR, Haenggeli C, Huang YH, Bergles DE, Jin L, Dykes Hoberg M, Vidensky S, Chung DS, Toan SV, Bruijn LI, Su ZZ, Gupta P, Fisher PB. Beta-lactam antibiotics offer neuroprotection by increasing glutamate transporter expression. Nature. 2005 Jan 6;433(7021):73-7. doi: 10.1038/nature03180. PMID 15635412
- [Background] Scahill L, Riddle MA, McSwiggin-Hardin M, Ort SI, King RA, Goodman WK, Cicchetti D, Leckman JF. Children's Yale-Brown Obsessive Compulsive Scale: reliability and validity. J Am Acad Child Adolesc Psychiatry. 1997 Jun;36(6):844-52. doi: 10.1097/00004583-199706000-00023. PMID 9183141
- [Background] Schafer JL, Graham JW. Missing data: our view of the state of the art. Psychol Methods. 2002 Jun;7(2):147-77. PMID 12090408
- [Background] Seber, G. A. F. Multivariate Observations. New York: Wiley, 1984.
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Shytle RD, Silver AA, Sheehan KH, Wilkinson BJ, Newman M, Sanberg PR, Sheehan D. The Tourette's Disorder Scale (TODS): development, reliability, and validity. Assessment. 2003 Sep;10(3):273-87. doi: 10.1177/1073191103255497. PMID 14503651
- [Background] Singer HS, Giuliano JD, Zimmerman AM, Walkup JT. Infection: a stimulus for tic disorders. Pediatr Neurol. 2000 May;22(5):380-3. doi: 10.1016/s0887-8994(00)00131-4. PMID 10913730
- [Background] Snider LA, Lougee L, Slattery M, Grant P, Swedo SE. Antibiotic prophylaxis with azithromycin or penicillin for childhood-onset neuropsychiatric disorders. Biol Psychiatry. 2005 Apr 1;57(7):788-92. doi: 10.1016/j.biopsych.2004.12.035. PMID 15820236
- [Background] Sorensen JL, Hargreaves WA, Friedlander S. Child global rating scales: selecting a measure of client functioning in a large mental health system. Eval Program Plann. 1982;5(4):337-47. doi: 10.1016/0149-7189(82)90006-4. PMID 10315340
- [Background] Storch EA, Geffken GR, Merlo LJ, Mann G, Duke D, Munson M, Adkins J, Grabill KM, Murphy TK, Goodman WK. Family-based cognitive-behavioral therapy for pediatric obsessive-compulsive disorder: comparison of intensive and weekly approaches. J Am Acad Child Adolesc Psychiatry. 2007 Apr;46(4):469-478. doi: 10.1097/chi.0b013e31803062e7. PMID 17420681
- [Background] Storch EA, Murphy TK, Geffken GR, Mann G, Adkins J, Merlo LJ, Duke D, Munson M, Swaine Z, Goodman WK. Cognitive-behavioral therapy for PANDAS-related obsessive-compulsive disorder: findings from a preliminary waitlist controlled open trial. J Am Acad Child Adolesc Psychiatry. 2006 Oct;45(10):1171-8. doi: 10.1097/01.chi.0000231973.43966.a0. PMID 17003662
- [Background] Storch EA, Murphy TK, Geffken GR, Sajid M, Allen P, Roberti JW, Goodman WK. Reliability and validity of the Yale Global Tic Severity Scale. Psychol Assess. 2005 Dec;17(4):486-91. doi: 10.1037/1040-3590.17.4.486. PMID 16393016
- [Background] Storch EA, Murphy TK, Geffken GR, Soto O, Sajid M, Allen P, Roberti JW, Killiany EM, Goodman WK. Further psychometric properties of the Tourette's Disorder Scale-Parent Rated version (TODS-PR). Child Psychiatry Hum Dev. 2004 Winter;35(2):107-20. doi: 10.1007/s10578-004-1880-7. PMID 15577277
- [Background] Swanson, J. M. School-based assessments and interventions for ADD students. Irvine, CA: K C Publishing, 1992.
- [Background] Swedo SE, Leonard HL, Garvey M, Mittleman B, Allen AJ, Perlmutter S, Lougee L, Dow S, Zamkoff J, Dubbert BK. Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections: clinical description of the first 50 cases. Am J Psychiatry. 1998 Feb;155(2):264-71. doi: 10.1176/ajp.155.2.264. PMID 9464208
- [Background] Tanner JM, Whitehouse RH. Clinical longitudinal standards for height, weight, height velocity, weight velocity, and stages of puberty. Arch Dis Child. 1976 Mar;51(3):170-9. doi: 10.1136/adc.51.3.170. PMID 952550
- [Background] Teixeira AL Jr, Guimaraes MM, Romano-Silva MA, Cardoso F. Serum from Sydenham's chorea patients modifies intracellular calcium levels in PC12 cells by a complement-independent mechanism. Mov Disord. 2005 Jul;20(7):843-5. doi: 10.1002/mds.20418. PMID 15747354
- [Background] Tuck MK, Chan DW, Chia D, Godwin AK, Grizzle WE, Krueger KE, Rom W, Sanda M, Sorbara L, Stass S, Wang W, Brenner DE. Standard operating procedures for serum and plasma collection: early detection research network consensus statement standard operating procedure integration working group. J Proteome Res. 2009 Jan;8(1):113-7. doi: 10.1021/pr800545q. PMID 19072545
- [Background] Tucker DM, Leckman JF, Scahill L, Wilf GE, LaCamera R, Cardona L, Cohen P, Heidmann S, Goldstein J, Judge J, Snyder E, Bult A, Peterson BS, King R, Lombroso P. A putative poststreptococcal case of OCD with chronic tic disorder, not otherwise specified. J Am Acad Child Adolesc Psychiatry. 1996 Dec;35(12):1684-91. doi: 10.1097/00004583-199612000-00022. PMID 8973076
- [Background] Wallwork B, Coman W, Mackay-Sim A, Greiff L, Cervin A. A double-blind, randomized, placebo-controlled trial of macrolide in the treatment of chronic rhinosinusitis. Laryngoscope. 2006 Feb;116(2):189-93. doi: 10.1097/01.mlg.0000191560.53555.08. PMID 16467702
- [Background] Wood, H. F., Feinstein, A. R., Taranta, A., & Simpson, R. Rheumatic fever in children and adolescents III. Comparative effectiveness of three prophylaxis regimens in preventing streptococcal infections and rheumatic fever. Annuals of Internal Medicine, 60(supplement 5), 31-46, 1964.
- [Background] Yamauchi K, Shibata Y, Kimura T, Abe S, Inoue S, Osaka D, Sato M, Igarashi A, Kubota I. Azithromycin suppresses interleukin-12p40 expression in lipopolysaccharide and interferon-gamma stimulated macrophages. Int J Biol Sci. 2009 Oct 23;5(7):667-78. doi: 10.7150/ijbs.5.667. PMID 19893639

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Participants consented to participate in the study. They completed baseline assessments but did not randomize to treatment.
Period: Overall Study
Arm/Group | Azithromycin | Placebo | Not Randomized
Started | 18 | 14 | 15
Completed | 18 | 14 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Participants only completed the baseline assessments but did not receive treatment.
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Not Randomized | Total
Number analyzed (Participants) | 18 | 14 | 15 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 14 | 15 | 47
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.78 (2.39) | 8.86 (3.11) | 7.21 (2.58) | 8.25 (2.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 9 | 21
  Male | 11 | 9 | 6 | 26
Region of Enrollment [Number; unit: participants]
  United States | 18 | 14 | 15 | 47

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: The CYBOCS is a clinician rated, semi-structured interview for rating the severity of OCD (Scahill, et al., 1997). Total scores range from 0 to 50, with higher scores representing greater severity. The total score is comprised of two subscores, obsessions and compulsions, each with a range of 0-25.
Time Frame: Before and after 4 week randomization
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 18 | 14
units on a scale
  Baseline | 29.49 (1.85) | 28.43 (2.04)
  After 4 week randomization | 20.53 (1.85) | 23.45 (2.09)

2. Secondary Outcome: Clinical Global Impressions-Severity OCD
Description: The CGI-S scale is a 7-point clinician rating of severity of psychopathology. Severity ratings range from 1 (no illness) to 7 (extremely severe). This instrument has been successfully used in treatment studies (Cook, et al., 2001; Storch, et al., 2007).
Time Frame: Before and after 4 week randomization
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Azithromycin | Placebo | Not Randomized
Number analyzed (Participants) | 18 | 14 | 0
units on a scale
  Baseline | 5.24 (0.23) | 5.00 (0.25) |
  After 4 week randomization | 4.06 (.23) | 4.93 (.25) |

3. Secondary Outcome: Screen for Childhood Anxiety-Related Emotional Disorders (SCARED)
Description: The Screen for Childhood Anxiety-Related Emotional Disorders (SCARED) is a 41-item parent and participant-completed tool used to measure symptoms of anxiety, including the most common symptoms of panic/somatic, generalized anxiety, separation anxiety, social phobia, and school phobia. Scores range from 0-82, with higher scores indicating more severe symptoms.The child and parent versions of the SCARED have moderate parent-child agreement and good internal consistency, test-retest reliability, and discriminant validity; it is also sensitive to treatment response (Birmaher et al. 1999). The target population for this rating is 8-18 years of age (Birmaher et al. 1997). The parent and child version of the SCARED were administered before and after week 4 randomization. This measure is not validated for use in 4-7 year olds.
Time Frame: Before and after 4 week randomization
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 18 | 14
units on a scale
  Baseline | 31.82 (3.75) | 20.43 (4.13)
  After 4 week randomization | 30.88 (3.75) | 21.97 (4.17)

ADVERSE EVENTS:
Time Frame: Before and after 4 week randomization
Groups:
- Azithromycin: This group was assigned to receive azithromycin (antibiotic).
- Placebo: This group was assigned to receive placebo (compound thickening agent with sugar and flavor additives - not active treatment).
Arm/Group | Azithromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 9/18 | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=18) | Placebo (N=14)
Loose stools (Gastrointestinal disorders) | 9 | 1
Constipation (Gastrointestinal disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No